CLINICAL TRIAL: NCT02640196
Title: A Comparison of Three Videolaryngoscopes for Double-lumen Tubes Intubation in Simulated Easy and Difficult Airways
Brief Title: Videolaryngoscopes for Double Lumen Tube Intubations in Simulated Easy and Difficult Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ANESTH-03-15
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Staff Anaesthesiologists; Limited Experience in Using Videolaryngoscopes
Keywords: Laryngoscope; Macintosh; Glidescope; King Vision; Airtraq; Double Lumen Tube

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Macintosh (Placebo Comparator): The participants intubated the easy airway simulator with a double lumen tube using the Macintosh laryngoscope followed with intubating the difficult airway simulator
  Interventions: Device: Macintosh
- GlideScope (Placebo Comparator): The participants intubated the easy airway simulator with a double lumen tube using the GlideScope laryngoscope followed with intubating the difficult airway simulator
  Interventions: Device: GlideScope
- Airtraq (Active Comparator): The participants intubated the easy airway simulator with a double lumen tube using the Airtraq laryngoscope followed with intubating the difficult airway simulator
  Interventions: Device: Airtraq
- King Vision (Active Comparator): The participants intubated the easy airway simulator with a double lumen tube using the King Vision followed with intubating the difficult airway simulator
  Interventions: Device: King Vision

INTERVENTIONS:
Device: Macintosh — The participants intubated the easy airway simulator with a double lumen tube using the Macintosh laryngoscope followed with intubating the difficult airway simulator
  Arms: Macintosh
Device: GlideScope — The participants intubated the easy airway simulator with a double lumen tube using the GlideScope followed with intubating the difficult airway simulator
  Arms: GlideScope
Device: Airtraq — The participants intubated the easy airway simulator with a double lumen tube using the Airtraq followed with intubating the difficult airway simulator
  Arms: Airtraq
Device: King Vision — The participants intubated the easy airway simulator with a double lumen tube using the King Vision followed with intubating the difficult airway simulator
  Arms: King Vision

SUMMARY:
The investigators hypothesized that the use of the King Vision™ and the Airtraq® VL would reduce the time to DLT intubation compared with the GlideScope® and Macintosh in simulated easy and difficult airways. The investigators have considered to assess the efficacy of each device in manikins before considering to evaluate them in patients undergoing thoracic procedures.

Twenty-one staff anaesthesiologists who had limited prior experience in using the VLs for DLT intubation participated in this randomised crossover study. Following a brief demonstration and two practice attempts, participants were volunteered to insert a DLT using the Macintosh, GlideScope®, Airtraq®, and King Vision™ on two high-fidelity easy and difficult airway simulators in a computer-generated randomized sequence. The primary endpoint, time to DLT intubation, as well as, the views obtained at laryngoscopy, ease of intubation, numbers of laryngoscopy attempts and optimisation manoeuvers, and failure to intubation; defined as an attempt took longer than 150 seconds, were recorded.

DETAILED DESCRIPTION:
Several regional surveys demonstrated that most thoracic anesthesiologists are using the double-lumen endobronchial tubes (DLT) as the first-choice lung separation technique. DLT, when compared with single lumen tracheal tube, can be more difficult to insert in patients with difficult airways. The videolaryngoscopes (VL) have the potential to facilitate the placement of the DLTs for lung separation in patients with predicted or unanticipated difficult airway.

The use of GlideScope® (Verathon Inc., Bothell, WA, USA), a VL with an angulated blade, has been associated with variable times to DLT intubation according to the prior experience of the operators, despite superior visualization of the glottis The channeled Airtraq® (Prodol Meditec S.A., Vizcaya, Spain) and standard non-channeled blade of the King Vision™ (Ambu, Ballerup, Copenhagen, Denmark), may offer additional benefits for DLT intubation in patients with limited mouth opening or restricted neck movement, in whom the use of traditional VL like as the Glidescope® could be difficult. This is because of the larger outer diameter, the distal curvature and the increased rigidity of the DLT. Of note, the longer times to DLT intubation with the use of different VL could be shortened with building up the operator's experience.

To the best of the investigators knowledge, the comparison of the effects of the Macintosh, GlideScope®, Airtraq®, and King Vision™ VL on the time to DLT intubation in simulated easy and difficult airways has not yet been studied.

Two high-fidelity simulators (Airway Management Trainer, model AA-3100, Laerdal, Kent, UK) were prepared to simulate easy and difficult airway situations, as described by Marshall et al. and Wang et al. The "easy" airway was established with the manikin in a neutral position. The "difficult" airway setting was obtained by placing an Oasis Elite™ Prone Head Rest, Adult (140 mm in height) (Covidien, Mansfield, MA) under the occiput and securing the head position with adhesive tape, object to replicate cervical-collar use. Positioning was confirmed after each attempt to ensure consistency.

ELIGIBILITY:
Inclusion Criteria:

* Staff anesthesiologists
* Signed consent
* Limited experience in using videolaryngoscopes for inserting double lumen tubes

Exclusion Criteria:

* Decline to sign the consent
* Non receiving the prior training demonstration
* Non practicing once with each device tested on each simulator scenario

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Time to achieve successful double lumen tube intubation | for 6 min after using each device
  defined as the time when the investigated laryngoscope passed the central incisors to when the tip of the bronchial lumen passed through the glottis, as confirmed visually by the operator (in the Macintosh group) or by the investigator, thanks to remote screens (in the VLs groups).

SECONDARY OUTCOMES:
Best view during laryngoscopy using the classification described by Cormack and Lehane | for 1 min after laryngoscopy
  using the classification described by Cormack and Lehane
Difficulty of intubation using a Visual Analog Scale (VAS) | for 6 min after using each device
  The difficulty of intubation was evaluated using a visual analog scale (VAS) (ranging from 0: extremely easy, to 100: extremely difficult) expressed by the anesthesiologists after the DLT intubation
Number of first-pass success | for 3 min after using each device
  first-pass success calculated as number of first-attempt successes/number of patients with an intubation attempt
Number of the required optimisation manoeuvers | for 6 min after using each device
  When the anaesthesiologists encountered difficulty in visualising vocal cords or placing the tube, they were allowed to use any manoeuver they would normally use to navigate the tube into the trachea including readjustment of the blade or tube or to ask the supervising investigator to help solve the problem, and gave suggestions or instructions

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, MD, Principal Investigator — Anesthesiology Department, Dammam University, Dammam, Saudi Arabia; Abdulmohsen A Al Ghamdi, MD, Study Director — Anesthesiology Department, Dammam University, Dammam, Saudi Arabia
Locations (1):
- Dammam University KFHU, Khobar, EP, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No